CLINICAL TRIAL: NCT03131141
Title: An Open Label, Single-dose, Single-period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of 14C-BC-3781 Administered Via the Intravenous or Oral Routes to Healthy Male Subjects
Brief Title: A Study to Assess Mass Balance Recovery, Metabolite Profile and Identification of IV and Oral 14C-BC-3781
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nabriva Therapeutics AG (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NAB-BC-3781-1013
Record Dates: First submitted 2017-02-16; First posted 2017-04-27 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Healthy
MeSH Terms: interventions — lefamulin

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Cohort A will receive a single IV administration of 14C-BC-3781 containing 150 mg BC-3781 and NMT 4.3 MBq (117 µCi) 14C, administered as an infusion over 60 min after a light breakfast
  Interventions: Drug: BC-3781
- Cohort B (Experimental): Cohort B will receive a single oral administration of 14C-BC-3781 containing 600 mg BC-3781 and NMT 4.1 MBq (112 µCi) 14C, in the fasted state
  Interventions: Drug: BC-3781

INTERVENTIONS:
Drug: BC-3781 — Lefamulin (BC-3781) is a potent, semi-synthetic antibacterial belonging to a novel class for systemic human use known as the pleuromutilins
  Other Names: Lefamulin

SUMMARY:
This is a single-centre, open-label, non-randomized, single dose study in healthy male subjects designed to assess mass balance recovery, metabolite profile and metabolite identification of radio-labeled BC-3781 administered via the intravenous or oral routes.

DETAILED DESCRIPTION:
This is a single-centre, open-label, non-randomised, single dose study to assess the pharmacokinetics, mass balance recovery, and metabolite profiling and identification following administration of iv or oral 14C-BC-3781 to healthy male subjects It is planned to enrol 2 cohorts of 5 subjects or 10 subjects in total. The active substance being investigated in this study is radiolabeled lefamulin ([14C] BC 3781), present in the investigational medicinal products (IMPs) as the acetate salt ([14C]-BC-3781.Ac).

Subjects assigned to Cohort A will receive a single IV administration of 14C-BC-3781 containing 150 mg BC-3781 and not more than (NMT) 4.3 MBq (117 µCi) 14C, administered as an infusion over 60 min after a light breakfast.

Subjects assigned to Cohort B will receive a single oral administration of 14C-BC-3781 containing 600 mg BC-3781 and NMT 4.1 MBq (112 µCi) 14C, in the fasted state

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Aged 30 to 65 years
* Body mass index of 18.0 to 35.0 kg/m2, inclusive
* Must have regular bowel movements
* Must provide written informed consent
* Must agree to use an adequate method of contraception

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the previous 3 months
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in males >21 units per week and females >14 units per week
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
* Subjects who have been dosed in an ADME study in the last 12 months
* Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator
* Positive drugs of abuse test result at screening and admission
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <90 mL/min using the Cockcroft-Gault equation
* Significant history of cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, or psychiatric disorders as judged by the investigator
* A familial history or presence of Long QT syndrome
* Subjects with QT interval corrected according to Fridericia's formula (QTcF) >480 ms
* A serum potassium level of less than 3.5 mmol/L at screening
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator.
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Have taken medications known to be strong P-gp inhibitors, or strong CYP3A4 inducers or inhibitors, within 28 days before IMP administration
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol or herbal remedies) in the 14 days before IMP administration

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2017-01-08 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Amount of radioactivity eliminated in urine | Day 1 pre-dose to Day 8 post-dose
  Amount excreted (Ae) and AE as a percentage of administered dose (%Ae)
Amount of radioactivity eliminated in feces | Day 1 pre-dose to Day 8 post-dose
  Amount excreted (Ae) and AE as a percentage of administered dose (%Ae)
Amount of radioactivity eliminated in urine and feces | Day 1 pre-dose to Day 8 post-dose
  Amount excreted (Ae) and AE as a percentage of administered dose (%Ae)
Cumulative amount of radioactivity eliminated in urine | Day 1 pre-dose to Day 8 post-dose
  Cumulative recovery (CumAe)and CumAe as a percentage of the dose (Cum%Ae)
Cumulative amount of radioactivity eliminated in feces | Day 1 pre-dose to Day 8 post-dose
  Cumulative recovery (CumAe)and CumAe as a percentage of the dose (Cum%Ae)
Cumulative amount of radioactivity eliminated in urine and feces | Day 1 pre-dose to Day 8 post-dose
  Cumulative recovery (CumAe)and CumAe as a percentage of the dose (Cum%Ae)

SECONDARY OUTCOMES:
Safety - hematology | Day 1 pre-dose to Day 8 post-dose
  Safety as assessed by review of changes in hematology
Safety - clinical chemistry | Day 1 pre-dose to Day 8 post-dose
  Safety as assessed by review of changes in clinical chemistry
Safety - urinalysis | Day 1 pre-dose to Day 8 post-dose
  Safety as assessed by review of changes in urinalysis
Safety - electrocardiograms | Day 1 pre-dose to Day 8 post-dose
  Safety as assessed by review of changes in electrocardiograms
Safety - vital signs | Day 1 pre-dose to Day 8 post-dose
  Safety as assessed by review of changes in vital signs
Safety - adverse events | Day 1 pre-dose to Day 8 post-dose
  Safety as assessed by review of adverse events
Metabolic profiling and structural identification in plasma | Day 1 pre-dose to Day 8 post-dose
  Number of metabolites >10% of circulating radioactivity in plasma
Metabolic profiling and structural identification in urine | Day 1 pre-dose to Day 8 post-dose
  Number of metabolites >10% of the dose in urine
Metabolic profiling and structural identification in feces | Day 1 pre-dose to Day 8 post-dose
  Number of metabolites >10% of the dose in feces
PK of total radioactivity: lag time (tlag), BC-3781 and major metabolites | Day 1 pre-dose to Day 8 post-dose
  Assessment of pharmacokinetics of lefamulin as assessed by radioactivity lag time
PK of total radioactivity: Cmax | Day 1 pre-dose to Day 8 post-dose
  Peak plasma concentration (Cmax), BC-3781 and major metabolites
PK of total radioactivity: AUC | Day 1 pre-dose to Day 8 post-dose
  area under the plasma concentration-time curve from time zero to time of last measurable concentration (AUC last) of BC-3781 and major metabolites
PK of total radioactivity: AUC (0-infinity) | Day 1 pre-dose to Day 8 post-dose
  area under the plasma concentration-time curve from time zero to infinity (AUCinf), BC-3781 and major metabolites
PK of total radioactivity: Time to Cmax | Day 1 pre-dose to Day 8 post-dose
  Time to reach total maximum observed concentration (tmax), BC-3781 and major metabolites
PK of total radioactivity: elimination half-life | Day 1 pre-dose to Day 8 post-dose
  elimination half-life (t1/2), BC-3781 and major metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Elyse Seltzer, MD, Study Director — Nabriva Therapeutics AG
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No